CLINICAL TRIAL: NCT03751982
Title: Improving Spatiotemporal Precision in Noninvasive Electrical Neuromodulation
Brief Title: Closed Loop TES for Enhancing Slow Wave Sleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brain Electrophysiology Laboratory Company (Industry)
Responsible Party: Principal Investigator, Don M. Tucker, CEO, Senior Scientist, Brain Electrophysiology Laboratory Company
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1R44MH115955 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Sleep Disturbance; Insomnia
Keywords: transcranial electrical stimulation
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Within subjects comparison of two effective treatments. Order of treatment is randomized and counterbalanced.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The phase alignment of the treatment is set in software and not revealed to participant or experimenter. Order of treatment is randomized and counterbalanced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-Loop (Active Comparator): In this arm of this repeated measures (within subjects) design, the participants receive electrical neuromodulation (TES) that is not synchronized to their slow waves of sleep. The Transcranial Electrical Stimulation (TES) is 2 mA applied in 100 ms pulses at 0.75 Hz.
  Interventions: Device: Transcranial Electrical Neuromodulation (TES)
- Closed-Loop (Experimental): In this arm of this repeated measures (within subjects) design, the participants receive electrical neuromodulation (TES) that is synchronized to their slow waves of sleep. The Transcranial Electrical Stimulation (TES) is 2 mA applied in 100 ms pulses at 0.75 Hz.
  Interventions: Device: Transcranial Electrical Neuromodulation (TES)

INTERVENTIONS:
Device: Transcranial Electrical Neuromodulation (TES) — TES phase-aligned with slow waves or not

SUMMARY:
Compare closed-loop with open-loop application of TES to enhance slow waves of sleep.

DETAILED DESCRIPTION:
Note: FDA has determined that TES with the stimulus parameters as specified for this trial presents no significant risk, so that FDA clearance is not required.

Several findings suggest that Transcranial Electrical Stimulation (TES) may be particularly effective if it is aligned with ongoing brain activity. One condition of the present research is an open-loop design, in which TES pulses (0.75 Hz pulses; 2.0 mA) are presented during slow wave sleep. The other condition is a closed-loop design, using identical pulses, but these will be phase aligned with the slow waves of sleep, measured by the electroencephalogram (EEG). The hypothesis is that closed-loop TES will be more effective in enhancing the amplitude and duration of slow wave sleep than open-loop TES.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* persons with epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-14 (Estimated); Primary Completion 2021-01-14 (Estimated); Study Completion 2022-01-14 (Estimated)

PRIMARY OUTCOMES:
Slow wave amplitude | Slow Wave Amplitude will be assessed during the night of sleep (defined as 8 hours). The dependent measure for the statistical test will be slow wave amplitude expressed per minute of stage N3 sleep for the study night.
  Amplitude of slow waves of sleep
Slow wave duration | Slow Wave Duration will be assessed in minutes for the night of sleep (defined as 8 hours). The dependent measure for the statistical test will be the duration (in minutes) of slow wave stage N3 sleep for the study night.
  Duration of slow wave period in sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Electrophysiology Laboratory Company, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No